CLINICAL TRIAL: NCT06944275
Title: Characterising the Loss of Haemostasis in Haemorrhagic Fever With Renal Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Institute of microbiology and immunology, Slovenia (Unknown)
Responsible Party: Sponsor
Other Study IDs: 25-011
Record Dates: First submitted 2025-02-13; First posted 2025-04-25 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Haemorrhagic Fever With Renal Syndrome
MeSH Terms: conditions — Hemorrhagic Fever with Renal Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples Without DNA — 2.5ml of blood will be collected in a PAXgene® Blood RNA Tube from each patient for the purposes of performing viral and host transcriptomic analysis. Following completion of sequencing analysis, remaining sample will be stored for use in future translation research relating to hantaviruses. Participants will be consented for the storage and future use of this sample.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-haemorrhagic cases: This cohort will include laboratory confirmed cases of haemorrhagic fever with renal syndrome without any evidence of haemorrhagic manifestations.
  Interventions: Procedure: Blood draw for thromboelastography - admission; Procedure: Blood draw for thromboelastography - follow-up; Procedure: Blood draw for transcriptomic analysis; Other: Data collection - clinical/demographic/epidemiological data; Other: Data collection - routine laboratory parameters; Other: Severity score calculation
- Haemorrhagic cases: This cohort will include laboratory confirmed cases of haemorrhagic fever with renal syndrome with evidence of haemorrhagic manifestations.
  Interventions: Procedure: Blood draw for thromboelastography - admission; Procedure: Blood draw for thromboelastography - follow-up; Procedure: Blood draw for transcriptomic analysis; Other: Data collection - clinical/demographic/epidemiological data; Other: Data collection - routine laboratory parameters; Other: Severity score calculation

INTERVENTIONS:
Procedure: Blood draw for thromboelastography - admission — Two blood samples will be collected at admission for thromboelastography using the TEG 6s platform (Haemonetics®). One sample will be collected in a citrated blood tube for global haemostasis assessment, and one sample will be collected in a heparinised tube for platelet function analysis.
Procedure: Blood draw for thromboelastography - follow-up — Two blood samples will be collected 3 - 7 days after initial thromboelastography for follow-up analysis using the TEG 6s platform (Haemonetics®). One sample will be collected in a citrated blood tube for global haemostasis assessment, and one sample will be collected in a heparinised tube for platelet function analysis.
Procedure: Blood draw for transcriptomic analysis — One blood sample will be collected at admission for transcriptomic analysis. Blood sample will be collected into a PAXgene® RNA tube and analysed using nanopore sequencing to characterise the viral and host transcriptome.
Other: Data collection - clinical/demographic/epidemiological data — Routine clinical/demographic/epidemiological data will be collected at admission and throughout hospitalisation. This will relate to clinical presentation (day of illness at presentation, presenting symptoms); demographics and epidemiology (age, gender, site of infection); clinical course during hospitalisation (maximum level of care, dialysis use, blood product use, survival outcome).
Other: Data collection - routine laboratory parameters — Data on routine laboratory parameters will be collected throughout hospitalisation. These will relate to laboratory clotting parameters (platelet count, prothrombin time, activated partial thromboplastin time, fibrinogen, D-dimer); liver function tests (aspartate aminotransferase, alanine aminotransferase); laboratory haematology parameters (haemoglobin, white cell count, blood film); laboratory biochemistry parameters (urea, creatinine); viral load.
Other: Severity score calculation — A severity score will be assigned to each patient based on clinical and laboratory data at admission according to a pre-defined scoring system.

SUMMARY:
Hantaviruses are globally distributed viruses that cause haemorrhagic fever with renal syndrome (HFRS) in Europe, a disease characterised by acute kidney failure and, in some cases, significant bleeding complications. The mechanisms underlying clotting abnormalities in HFRS remain poorly understood. This study aims to investigate the pathological mechanisms of clotting dysfunction in hospitalised HFRS patients, assess the impact of different hantavirus types on disease severity, and evaluate the accuracy of a severity scoring system developed in China for predicting mortality in European patients.

Hospitalised patients with laboratory-confirmed HFRS will be prospectively recruited from University Medical Centre Ljubljana, Slovenia. Blood samples will be analysed for routine laboratory markers, thromboelastography (TEG) will assess real-time clotting function, and transcriptomic analysis will identify hantavirus strains and gene expression patterns linked to disease severity. Patients will be stratified into haemorrhagic and non-haemorrhagic groups, with statistical analyses comparing clinical and laboratory parameters to identify predictors of bleeding risk. Findings from this study may contribute to improved risk stratification and potential therapeutic targets for HFRS.

DETAILED DESCRIPTION:
Hantaviruses are globally distributed viruses that are transmitted to humans through the inhalation of viral particles found in the urine and faeces of infected rodents. In Europe, hantaviruses cause haemorrhagic fever with renal syndrome (HFRS), a disease characterised by acute kidney failure and, in some cases, significant bleeding complications. Despite advances in understanding HFRS, the mechanisms underlying these bleeding abnormalities remain poorly understood. Several hypotheses suggest that hantaviruses may interfere with the function of blood clotting factors, but definitive evidence is lacking.

Slovenia, a country in southern Europe, has one of the highest incidences of HFRS relative to its population, with recent years seeing large outbreaks. Discussions with leading hantavirus experts in Slovenia have highlighted the urgent need for further research, particularly to understand why some patients with HFRS develop severe bleeding complications. Currently, no licensed treatments exist for HFRS, raising concerns about future outbreaks, which are expected to become more frequent due to climate change. By investigating the mechanisms leading to clotting dysfunction, this study aims to identify potential targets for future therapeutic interventions.

This study will explore the pathological mechanisms driving clotting abnormalities and bleeding in hospitalised patients with HFRS. Additionally, it will assess whether different hantavirus types influence disease severity and haemorrhagic complications and evaluate the applicability of a severity scoring system-originally developed for HFRS cases in China-in predicting outcomes among Slovenian patients.

Patients with laboratory-confirmed HFRS will be prospectively recruited from University Medical Centre Ljubljana, Slovenia. Blood samples will be collected at multiple time points during their illness and tested for standard laboratory markers, including clotting factors, blood cell counts, kidney function, and liver function. Additionally, thromboelastography (TEG) will be performed to assess real-time clotting dynamics, providing a more detailed evaluation of clotting abnormalities.

An additional blood sample will undergo transcriptomic analysis using nanopore sequencing. This will identify the specific hantavirus strain in each patient and analyse gene expression patterns associated with disease severity and bleeding risk. Patients will also be assigned a severity score based on their clinical presentation, laboratory results, and symptoms, using a scoring system developed in China to predict HFRS-related mortality. This study will evaluate the reliability of this scoring system in a European cohort.

To better understand the factors contributing to bleeding in HFRS, patients will be categorised into two groups: those with haemorrhagic manifestations and those without. Statistical analyses will compare laboratory and clinical findings between these groups, aiming to identify key predictors of bleeding complications. The findings from this research may help inform future therapeutic strategies for HFRS.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older, including pregnant women
* Laboratory-confirmed HFRS (serology and/or RT-PCR)
* Willing and able to provide informed consent

Exclusion Criteria:

* Patients under 18 years of age
* Co-infections with other pathogens
* Pre-existing coagulation disorders
* Use of anticoagulant medication
* Inability or refusal to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the University Medical Centre Ljubljana. Suspected cases of HFRS will be identified based on a clinical case definition of presence of fever and one of the following: acute kidney injury (AKI), thrombocytopenia, bleeding, or epidemiological risk. Cases will be confirmed for inclusion in the study following laboratory confirmation of hantavirus infection using serological methods for antibody detection or reverse transcription polymerase chain reaction (RT-PCR) to detect hantavirus genetic material in the blood.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Reaction Time (R) on thromboelastography from admission to follow-up (3-7 days), assessing clot initiation and its association with haemostatic dysfunction in HFRS. | Baseline and 3-7 days later
  Reaction time (R): The amount of time between the start of the test and the beginning of coagulation. Measured in minutes (min). Measured according to standardised assay on the TEG 6s haemostasis analyser.
Change in K-Time (K) on thromboelastography from admission to follow-up (3-7 days), evaluating clot kinetics and fibrin polymerisation in relation to haemostatic abnormalities in HFRS. | Baseline and 3-7 days later
  K-time (K): The speed of formation of the clot from Reaction Time (R) to a specific clot strength. Measured in minutes (min). Measured according to standardised assay on the TEG 6s haemostasis analyser.
Change in Alpha Angle (α-Angle) on thromboelastography from admission to follow-up (3-7 days), reflecting fibrin build-up and clot formation rate in patients with HFRS. | Baseline and 3-7 days later
  Alpha Angle (α-Angle): The speed of clot strengthening. Measured in degrees (°). Measured according to standardised assay on the TEG 6s haemostasis analyser.
Change in Maximum Amplitude (MA) on thromboelastography from admission to follow-up (3-7 days), assessing overall clot strength and platelet contribution to clot stability in HFRS. | Baseline and 3-7 days later
  Maximum Amplitude (MA): The ultimate strength of the clot. Measured in millimetres (mm). Measured according to standardised assay on the TEG 6s haemostasis analyser.
Change in Lysis 30 (LY30) on thromboelastography from admission to follow-up (3-7 days), measuring fibrinolysis and clot breakdown in relation to bleeding risk in HFRS. | Baseline and 3-7 days later
  Lysis 30 (LY30): Percent lysis 30 minutes after Maximum Amplitude (MA) is finalised. The LY30 measurement is based on the reduction of the tracing area that occurs between the time that MA is measured until 30 minutes after the MA is finalised. Measured as a percentage (%). Measured according to standardised assay on the TEG 6s haemostasis analyser.
Change in Percentage Inhibition (% Inhibition) on thromboelastography from admission to follow-up (3-7 days), evaluating the effect of antithrombotic pathways on clot formation in HFRS. | Baseline and 3-7 days later
  Percentage Inhibition (% Inhibition): Indicates the reduction in platelet contribution to overall clot strength. Measured as a percentage (%). Measured according to standardised assay on the TEG 6s haemostasis analyser.
Change in Percentage Aggregation (% Aggregation) on thromboelastography from admission to follow-up (3-7 days), assessing platelet function and its role in haemostatic dysfunction in HFRS. | Baseline and 3-7 days later
  Percentage Aggregation (% Aggregation): Indicates the percent of platelets not inhibited, determined by comparing the uninhibited platelet contribution to the baseline platelet contribution. Measured as a percentage (%). Measured according to standardised assay on the TEG 6s haemostasis analyser.

SECONDARY OUTCOMES:
Change in platelet count over the course of illness, assessing thrombocytopenia and its role in haemostatic dysfunction in HFRS. | Baseline (day 1) and daily thereafter through hospitalisation, up to 21 days
  Platelet count measures the number of platelets in the blood, which are essential for clot formation. Measured as ×10⁹/L. Change over the course of illness, measured in days.
Change in prothrombin time (PT) over the course of illness, evaluating coagulation factor activity and clotting dysfunction in HFRS. | Baseline (day 1) and daily thereafter through hospitalisation, up to 21 days
  Prothrombin time (PT) measures the time taken for blood to clot via the extrinsic pathway. Measured in seconds (s). Change over the course of illness, measured in days.
Change in activated partial thromboplastin time (APTT) over the course of illness, assessing abnormalities in the intrinsic clotting pathway in HFRS. | Baseline (day 1) and daily thereafter through hospitalisation, up to 21 days
  Activated partial thromboplastin time (APTT) assesses the intrinsic clotting pathway and measures time to clot formation. Measured in seconds (s). Change over the course of illness, measured in days.
Change in fibrinogen levels over the course of illness, investigating fibrinogen consumption and clot formation abnormalities in HFRS. | Baseline (day 1) and daily thereafter through hospitalisation, up to 21 days
  Fibrinogen is part of clotting assessment and is a key protein involved in clot formation, converted into fibrin to stabilise clots. Measured in g/L. Change over the course of illness, measured in days.
Change in D-dimer levels over the course of illness, evaluating fibrinolysis and its association with haemorrhagic complications in HFRS | Baseline (day 1) and daily thereafter through hospitalisation, up to 21 days
  D-dimer is a marker of fibrin breakdown, used to assess fibrinolysis and clotting activity. Measured in ng/mL. Change over the course of illness, measured in days.
Change in aspartate aminotransferase (AST) over the course of illness, assessing liver involvement and potential contributions to haemostatic dysfunction in HFRS. | Baseline (day 1) and daily thereafter through hospitalisation, up to 21 days
  Aspartate aminotransferase (AST) is an enzyme released from damaged liver cells, used to assess liver injury. Measured in U/L. Change over the course of illness, measured in days.
Change in alanine aminotransferase (ALT) over the course of illness, evaluating liver injury and its association with disease severity in HFRS. | Baseline (day 1) and daily thereafter through hospitalisation, up to 21 days
  Alanine aminotransferase (ALT) is an enzyme released from damaged liver cells, used to assess liver injury. Measured in U/L. Change over the course of illness, measured in days.
Change in haemoglobin levels over the course of illness, assessing anaemia and its potential link to bleeding severity in HFRS. | Baseline (day 1) and daily thereafter through hospitalisation, up to 21 days
  Haemoglobin (Hb) measures the oxygen-carrying protein in red blood cells. Measured in g/L. Change over the course of illness, measured in days.
Change in white cell count (WCC) over the course of illness, evaluating immune response and its association with disease severity in HFRS. | Baseline (day 1) and daily thereafter through hospitalisation, up to 21 days
  White cell count (WCC) reflects the number of white blood cells, indicating immune response or infection. Measured in ×10⁹/L. Change over the course of illness, measured in days.
Change in blood film findings over the course of illness, identifying morphological changes in blood cells associated with HFRS severity. | Baseline (day 1) and daily thereafter through hospitalisation, up to 21 days
  A blood film is a microscopic evaluation of blood cells to assess morphology and detect abnormalities. This is a descriptive report with no numerical value. Change over the course of illness, measured in days.
Change in creatinine levels over the course of illness, evaluating renal impairment and disease progression in HFRS. | Baseline (day 1) and daily thereafter through hospitalisation, up to 21 days
  Creatinine is a marker of renal function, indicating kidney filtration efficiency. Measured in µmol/L. Change over the course of illness, measured in days.
Change in urea levels over the course of illness, assessing kidney dysfunction and its relationship to HFRS severity. | Baseline (day 1) and daily thereafter through hospitalisation, up to 21 days
  Urea is a waste product of protein metabolism, used to assess kidney function. Measured in mmol/L. Change over the course of illness, measured in days.
Day of illness at hospital presentation, assessing timing of medical intervention in relation to disease progression. | Baseline (at admission)
  The number of days of illness experienced prior to presentation to hospital, inclusive of day of presentation.
Frequency of symptoms at presentation and throughout hospitalisation, characterising the clinical course and severity of HFRS. | Baseline (day 1) and daily thereafter through hospitalisation, up to 21 days
  The occurrence and frequency of key symptoms (such as fever, bleeding, or kidney dysfunction) at the time of hospital presentation and during the hospital stay, used to characterise the clinical course and severity of HFRS.
Maximum level of clinical care required during hospitalisation, assessing disease severity and need for intensive care in HFRS patients. | Baseline (day 1) and daily thereafter through hospitalisation, up to 21 days
  The highest level of medical care required by the patient during their hospitalisation (e.g., general ward, high-dependency unit, or intensive care unit), used to assess disease severity and the need for intensive care in HFRS patients.
Survival outcome, evaluating overall mortality and predictors of fatal HFRS cases. | Baseline (day 1) and daily thereafter through hospitalisation, up to 21 days
  Outcome of each illness, recorded as either 'survival' or 'death'. Outcomes will only be observed from the point of illness onset until discharge from hospital.
Frequency of blood product use during hospitalisation, assessing transfusion requirements as a marker of haemorrhagic severity in HFRS. | Baseline (day 1) and daily thereafter through hospitalisation, up to 21 days
  The number of patients receiving blood products during hospitalisation. A blood product refers to any therapeutic component derived from human blood, including red blood cells, platelets, plasma, and clotting factor concentrates, used for transfusion or treatment of coagulation disorders.
Frequency of acute renal replacement therapy use during hospitalisation, evaluating the need for dialysis as an indicator of severe renal dysfunction in HFRS. | Baseline (day 1) and daily thereafter through hospitalisation, up to 21 days
  Number of patients requiring acute renal replacement therapy (RRT) during hospitalisation. Acute RRT refers to short-term treatments used to support kidney function in patients with acute kidney injury (AKI), including haemodialysis, haemofiltration, or continuous renal replacement therapy (CRRT), to remove waste products, excess fluids, and toxins from the blood.
Viral RNA genomic analysis and its association with disease severity and haemostatic dysfunction | Baseline (at admission)
  Nanopore sequencing of hantavirus RNA to identify the specific hantavirus strain present, using blood samples collected at the time of hospital admission. This will help determine if certain hantavirus strains are associated with more severe disease and increased haemostatic dysfunction in patients with HFRS.
Host RNA genomic analysis and its association with disease severity and haemostatic dysfunction | Baseline (at admission)
  Nanopore sequencing of host RNA to identify differentially expressed genes between cohorts, using blood samples collected at the time of hospital admission. This analysis will help investigate any host genetic factors that may be linked to disease severity and haemostatic dysfunction in patients with HFRS.
Validation of a severity score for predicting risk of death from HFRS in European patients | Baseline (at admission)
  Each patient will be assigned a severity score upon admission based on a scoring system developed by researchers in China, designed to predict the risk of death from HFRS. Each patient will be assigned a score of 0 - 22 according to the published scoring matrix. Scores of 0 - 10 are categorised as 'Low Risk'; scores of 11 - 14 are categorised as 'Medium Risk'; scores of 15 - 22 are categorised as 'High Risk'. The score will be calculated at baseline and then assessed for its correlation with the disease outcome (survival vs. death) to determine if it is applicable for use in European patients with HFRS.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hu H, Zhan J, Chen W, Yang Y, Jiang H, Zheng X, Li J, Hu F, Yu D, Li J, Yang X, Zhang Y, Wang X, Bi Z, Liang Y, Shen H, Du H, Lian J. Development and validation of a novel death risk stratification scale in patients with hemorrhagic fever with renal syndrome: a 14-year ambispective cohort study. Clin Microbiol Infect. 2024 Mar;30(3):387-394. doi: 10.1016/j.cmi.2023.11.003. Epub 2023 Nov 11. PMID 37952580